CLINICAL TRIAL: NCT02280096
Title: Efficacy and Safety of 4-aminopyridine on Cognitive Performance and Motor Function of Patients With Multiple Sclerosis. Randomized, Blinded, Placebo-controlled Clinical Trial.
Brief Title: Efficacy and Safety of 4-aminopyridine on Cognitive Performance and Motor Function of Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-785-091
Record Dates: First submitted 2014-10-10; First posted 2014-10-31 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive function; Multiple sclerosis; 4-aminopyridine; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — 4-Aminopyridine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4-aminopyridine treatment (Active Comparator): 4-aminopyridine is given as gelatin capsules containing 4-aminopyridine 10 mg and microcrystalline cellulose as the excipient. Each patient will take two capsules every 8 hours after meals, for a total of 6 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
  Interventions: Drug: 4-aminopyridine
- Placebo (Placebo Comparator): Patients randomized to the placebo sequence will receive placebo for 20 weeks after the run-in period. They will be blinded to the fact that they are taking placebo, and capsules will be identical in appearance to the intervention capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4-aminopyridine — Each patient will take two capsules every 8 hours after meals, for a total of 6 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
  Other Names: 4-AP
  Arms: 4-aminopyridine treatment
Drug: Placebo — The placebo arm will include Microcrystalline Cellulose placebo
  Other Names: Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
Twenty four relapsing-remitting multiple sclerosis (RRMS) patients over the age of 18, with similar degree of disability, and with an evolution of at last 6 months, who are in first-line immunomodulatory therapy and have a stable disease (no more than one outbreak per year) will be included in the present study. Patients will be administered a neuropsychological test battery selected for this study and divided into two sessions of one and a half-hour each. Emotional state will be assessed with the Beck Depression Inventory in a different session. Cognitive impairment is defined as the alteration of two or more neuropsychological tests. Patients will be divided randomly into two groups where one will receive placebo and the other one 4-Aminopyridine (4-AP) for a period of 22 weeks in increasing doses.

DETAILED DESCRIPTION:
Consecutive patients with stable multiple sclerosis are being recruited from the neurological services of Social Security Mexican Institute (IMSS) at the National Medical Center (CMN) "Siglo XXI" Specialties Hospital over the period of 1 year. Of those meeting inclusion criteria, 24 will be selected for the study. After signing an informed consent, they will be randomized into 12 for the intervention arm and 12 for the placebo arm. All patients will receive capsules for daily consumption according to their assignment, with no visible difference between capsules. Dosage will be 6.5-7.5 mg/kg to a limit of 50 mg. These capsules will be taken for a period of 22 weeks. A battery of neuropsychological tests will be administered at baseline, after 22 weeks, and after an additional 22 weeks of follow-up to assess cognitive performance and motor function. Emotional state will be assessed with the Beck Depression Inventory at each of the three afore mentioned points.

After the follow-up period, all test results will be analyzed and compared to determine the efficacy and safety of 4-aminopyridine on the cognitive performance and motor function of patients. Mann-Whitney U will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria: Patients with multiple sclerosis (MS) are eligible for the study if they meet the following criteria:

1. Relapsing recurrent MS with an evolution of at last 6 months before the study began.
2. Both males and females, aged 20 - 65 years
3. Neurologic Expanded Disability Status Scale (EDSS) 3 - 7
4. Who are in first-line immunomodulatory therapy and have a stable disease
5. No more than one outbreak per year.
6. The absence of antiepileptic antecedent and electroencephalogram without epileptic activity.
7. For females: postmenopausal or surgically sterile, or using an acceptable method of birth control

Exclusion Criteria:

1. History of cardiovascular disease (syncope, arrhythmia, or myocardial infarction within the last two years), systolic blood pressure greater than 150 or less than 70 mm Hg, diastolic blood pressure greater than 110 or less than 50 mm Hg, or heart rate greater than 110 or less than 50 beats/minute; impaired hepatic function (total hepatic enzyme or bilirubin levels greater than 2 times the upper limits of normal) or impaired renal function (creatinine level greater than 2 times the upper limits of normal) less than 6 months before the study
2. Known allergy to pyridine-containing drugs
3. Neurologic, degenerative, or psychiatric disorders that would impair the patient's ability to complete the protocol
4. Any illness or abnormality that would jeopardize patient safety or interfere with the conduct of the study
5. History of substance abuse
6. Inability to discontinue excluded concomitant drug therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Arreola Mora, MS, Principal Investigator — Instituto Mexicano del Seguro Social; Israel Grijalva, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Especialidades, CMN Siglo XXI, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruck T, Bittner S, Simon OJ, Gobel K, Wiendl H, Schilling M, Meuth SG. Long-term effects of dalfampridine in patients with multiple sclerosis. J Neurol Sci. 2014 Feb 15;337(1-2):18-24. doi: 10.1016/j.jns.2013.11.011. Epub 2013 Nov 16. PMID 24290498
- [Background] Amato MP, Portaccio E, Zipoli V. Are there protective treatments for cognitive decline in MS? J Neurol Sci. 2006 Jun 15;245(1-2):183-6. doi: 10.1016/j.jns.2005.07.017. Epub 2006 Apr 27. PMID 16643949
- [Background] Romani A, Bergamaschi R, Candeloro E, Alfonsi E, Callieco R, Cosi V. Fatigue in multiple sclerosis: multidimensional assessment and response to symptomatic treatment. Mult Scler. 2004 Aug;10(4):462-8. doi: 10.1191/1352458504ms1051oa. PMID 15327047
- [Background] Rossini PM, Pasqualetti P, Pozzilli C, Grasso MG, Millefiorini E, Graceffa A, Carlesimo GA, Zibellini G, Caltagirone C. Fatigue in progressive multiple sclerosis: results of a randomized, double-blind, placebo-controlled, crossover trial of oral 4-aminopyridine. Mult Scler. 2001 Dec;7(6):354-8. doi: 10.1177/135245850100700602. PMID 11795455
- [Background] Smits RC, Emmen HH, Bertelsmann FW, Kulig BM, van Loenen AC, Polman CH. The effects of 4-aminopyridine on cognitive function in patients with multiple sclerosis: a pilot study. Neurology. 1994 Sep;44(9):1701-5. doi: 10.1212/wnl.44.9.1701. PMID 7936300
- [Derived] Arreola-Mora C, Silva-Pereyra J, Fernandez T, Paredes-Cruz M, Bertado-Cortes B, Grijalva I. Effects of 4-aminopyridine on attention and executive functions of patients with multiple sclerosis: Randomized, double-blind, placebo-controlled clinical trial. Preliminary report. Mult Scler Relat Disord. 2019 Feb;28:117-124. doi: 10.1016/j.msard.2018.12.026. Epub 2018 Dec 19. PMID 30593980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four patients were recruited, of whom 21 completed the study
Pre-assignment Details: Three patients were excluded: one because of lack of adherence to the treatment; another presented an anxiety crisis and third one due to pregnancy. In the end, 11 patients were included in the treatment group and 10 in the placebo (control) group.
Groups:
- 4-aminopyridine Treatment: 4-aminopyridine is given as gelatin capsules containing 4-aminopyridine 10 mg and microcrystalline cellulose as the excipient. Each patient will take two capsules every 6 hours after meals, for a total of 6 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
  4-aminopyridine: Each patient will take two capsules every 6 hours after meals, for a total of 6 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
Period: Overall Study
Arm/Group | 4-aminopyridine Treatment | Placebo
Started | 13 | 11
Completed | 11 | 10
Not Completed | 2 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Functional neurological disorder | 1 | 0
Not completed — Lack of attachment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 4-aminopyridine Treatment (20 Weeks): 4-aminopyridine is given as gelatin capsules containing 4-aminopyridine 10 mg and microcrystalline cellulose as the excipient. Each patient will take two capsules every 8 hours after meals, for a total of 6 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
- Placebo (20 Weeks): Patients randomized to the placebo sequence will receive placebo for 20 weeks after the run-in period. They will be blinded to the fact that they are taking placebo, and capsules will be identical in appearance to the intervention capsules.
  Placebo: The placebo arm will include Microcrystalline Cellulose placebo
- Total: Total of all reporting groups
Arm/Group | 4-aminopyridine Treatment (20 Weeks) | Placebo (20 Weeks) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (8) | 34.3 (9.8) | 36.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 4 | 4 | 8
Weight [Mean (Standard Deviation); unit: kg] | 66.1 (18.3) | 76.1 (18.1) | 71.1 (18.2)
Disease duration [Mean (Full Range); unit: years] | 8.55 [2 to 20] | 9.4 [2 to 23] | 8.97 [2 to 23]
Education [Mean (Full Range); unit: years] | 15.9 [9 to 19] | 16.9 [10 to 24] | 16.4 [9 to 24]
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — It is a tool that can be used to assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The minimum score is 0 and the maximum score is 30. The cut-off point accepted as an indicator of cognitive decline is 23 or less. There are three levels of impairment: 0-17 severe cognitive impairment, 18-23 moderate and 24-30 without cognitive impairment.
  units on a scale | 27.1 (1.4) | 27 (1.6) | 27.05 (1.5)
Interferon beta 1a [Count of Participants; unit: Participants] | 1 | 2 | 3
Interferon beta 1b [Count of Participants; unit: Participants] | 6 | 4 | 10
Interferon beta 1a subcutaneous [Count of Participants; unit: Participants] | 3 | 2 | 5
Glatiramer acetate [Count of Participants; unit: Participants] | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Brief Repeatable Battery of Rao
Description: Neuropsychological tests to assess: verbal fluency. Participants have to say as many words as possible from a category in a given time 60 Sec (F, A, S) Max score 72 and min score 19 words. Higher scores indicate a better cognitive performance.
Time Frame: 10-15 minutes
Population: Word List Generation (3 trials/60 sec)
Measure: Mean (Standard Deviation); unit: Correct words
Groups:
- 4-aminopyridine: The mean dose provided to the patients was 0.63 ± 0.05 mg per kg of body weight.
- Placebo: Identical placebo capsules administered for 22 weeks.
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
Correct words | 42.09 (14.5) | 35.5 (6.6)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Test type: Superiority; p = 0.028, t-test, 1 sided; t-boostrap = 0.028

2. Primary Outcome: Integrated Program of Neuropsychological Exploration Test Barcelona
Description: Integrated Program of Neuropsychological Exploration Test Barcelona: Digit Span Forward (DSF), (attention spam and improved scoring metrics significantly enhance the precision of DSF assessments of short-term verbal memory). Digit sequences are presented beginning with a length of two digits and two trials are presented at each increasing list length. Max score 8 and min score 0 digits. Higher scores indicate a better cognitive performance.
Time Frame: 7-10 min
Population: Attention spam.
Measure: Mean (Standard Deviation); unit: correct numbers recalled
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
correct numbers recalled | 6.1 (1.5) | 5 (0.8)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Test type: Superiority; p = 0.001, t-test, 1 sided; t-boostrap = 0.001

3. Primary Outcome: Rey-Osterrieth Complex Figure Test (ROCF)
Description: The purpose of this test is to assess visual-spatial constructional ability and visual memory. The time required to copy the drawing is recorded. Less time indicates a better performance and more time indicates a worse outcome (min score 60 and max score 300 seconds).
Time Frame: 10-15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale (seconds)
Groups:
- 4-aminopyridine: The dose provided to the patients was 0.63 ± 0.05 mg per kg of body weight.
- Placebo: Identical placebo capsules were administered
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale (seconds) | 208.6 (121.2) | 231.2 (114.8)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Test type: Superiority; p = 0.016, t-test, 1 sided; t-boostrap = 0.016

4. Primary Outcome: Five Digit Test (FDT). Processing Speed
Description: Processing speed information (which includes reading, count, and alternation speed). Cards with a different number of stimuli are shown to the patient, who has to read, count, and respond to a change of instructions (alternation). Reading speed (min 12, max 31+ seconds), counting speed (min 14, max 28+ seconds), and alternation speed (min 26, max 56+ seconds) are recorded. Less speed corresponds to a better outcome.
Time Frame: 8-10 min
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- 4-aminopirydine: The mean dose provided to the patients was 0.63 ± 0.05 mg per kg of body weight.
Arm/Group | 4-aminopirydine | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Reading speed | 28 (9) | 29.6 (4.2)
  Count speed | 30.5 (9.2) | 34.2 (12)
  Alternation speed | 60.3 (25.7) | 58.8 (17.7)
Statistical Analysis 1: Comparison: 4-aminopirydine vs Placebo; Reading speed; Test type: Superiority; p = 0.64, t-test, 1 sided; t-boostrap = 0.64
Statistical Analysis 2: Comparison: 4-aminopirydine vs Placebo; Count speed; Test type: Superiority; p = 0.43, t-test, 1 sided; t-boostrap = 0.43
Statistical Analysis 3: Comparison: 4-aminopirydine vs Placebo; Alternation; Test type: Superiority; p = 0.9, t-test, 1 sided; t-boostrap = 0.9

5. Primary Outcome: Wisconsin Card Sorting Test (WCST)
Description: Is used primarily to assess perseveration and abstract thinking, allows the clinician to assess the following 'frontal' lobe functions: strategic planning, organised searching, utilising environmental feedback to shift cognitive sets, directing behaviour toward achieving a goal. WCST measures abstract reasoning and ability to alter problem solving strategies. Patients are given 128 response cards and 4 stimulus cards and asked to match each stimulus card to 1 pile of response cards. The patient is not told how to match the cards, only "right" or "wrong" to each placement. The examiner may change matching rules during the test. Perseveration errors occur when subject repeats the same error no matter how many times they are told the placement is wrong. Higher scores indicate a worse cognitive performance (min=0-3, max=58-126)
Time Frame: 10-15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | 19.8 (35.6) | 22.8 (32.2)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Test type: Superiority; p = 0.83, t-test, 1 sided; t-boostrap = 0.83

6. Primary Outcome: Color Trails Test (CTT)
Description: Measure sustained attention. The CTT uses numbered coloured circles and universal sign language symbols. The circles are printed with vivid pink or yellow backgrounds that are perceptible to colourblind individuals. For the Colour Trails 1 trial, the respondent uses a pencil to rapidly connect circles numbered 1 through 25 in sequence. Less time indicates better performance (min=10, max= 240).
Time Frame: 5-8 minutes
Population: Color Trails Test 1. Execution time
Measure: Mean (Standard Deviation); unit: units on a scale (seconds)
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale (seconds) | 68.91 (40.7) | 67.3 (37.4)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Test type: Superiority; p = 0.92, t-test, 1 sided; t-boostrap = 0.92

7. Primary Outcome: Tower Of London (TOL). Total Moves and Total Correct Moves
Description: Measures higher order problem-solving ability. The information it provides is not only useful when assessing frontal lobe damage, but also when evaluating attention disorders and executive functioning difficulties. The administrator arranges red, green, and blue beads on a peg board to match the configuration in the diagram. The patient is asked to replicate the configuration on a second peg board. Scores are calculated for Total Correct Moves and Total Moves. Total moves: higher scores indicate a worse cognitive performance (min= 0, max=58+); Total correct higher scores indicate a better cognitive performance (min=0, max=10).
Time Frame: 25-30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Total moves | 42.7 (19.7) | 50.8 (23.9)
  Correct moves | 4 (2.7) | 3 (1.9)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Total moves; Test type: Superiority; p = 0.017, t-test, 1 sided; t-boostrap = 0.017
Statistical Analysis 2: Comparison: 4-aminopyridine vs Placebo; Correct moves; Test type: Superiority; p = 0.010, t-test, 1 sided; t-boostrap = 0.010

8. Primary Outcome: Tower Of London (TOL). Execution Time and Problem-solving Time
Description: Measures higher-order problem-solving ability. The information it provides is not only useful when assessing frontal lobe damage, but also when evaluating attention disorders and executive functioning difficulties. The administrator arranges red, green, and blue beads on a peg board to match the configuration in the diagram. The patient is asked to replicate the configuration on a second peg board. Scores are calculated for Total Execution Time (since the patient performs the first move until he ends the test), Total Problem-Solving Time (the sum of planning and execution times). Total execution time higher scores indicate a worse outcome (min= 0-78, max=564+ seconds), Total problem-solving time higher scores indicate a worse outcome (min= 0-56, max=500+ seconds).
Time Frame: 25-30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Total execution time | 296.2 (109.3) | 367.9 (265.4)
  Total problem-solving time | 363.3 (130) | 426.8 (278.9)
Statistical Analysis 1: Comparison: 4-aminopyridine vs Placebo; Execution time; Test type: Superiority; p = 0.001, t-test, 1 sided; t-boostrap = 0.001
Statistical Analysis 2: Comparison: 4-aminopyridine vs Placebo; Problem-solving time; Test type: Superiority; p = 0.001, t-test, 1 sided; t-boostrap = 0.001

9. Secondary Outcome: Improved Physical Capacity
Description: The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. The first levels 1.0 to 4.5 refers to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refers to the loss of ambulatory ability. It also provides eight subscale measurements called Functional System (FS) scores. The levels of function within each category refer to the eight FS affected by MS: The FS are scored on a scale of 0 (low level of problems) to 5 (high level of problems) to best reflect the level of disability observed clinically.
Time Frame: 15-20 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-aminopyridine Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | 4.6 (1.55) | 4.04 (1.27)

10. Secondary Outcome: Fatigue
Description: The Fatigue Severity Scale (FSS) is one of the most frequently used inventories for measuring fatigue in people with chronic illnesses. The FSS questionnaire is comprised of nine statements inquiring about the examinee's sleep habits over the preceding week. Ratings are on a 7-point Likert scale, where higher scores indicate how strongly the patient agrees with the nine statements.Scale. Scoring using a bimodal response system or a Likert score with weights assigned to each response choice. Likert or bimodal rating scales with 4 response options. For the Likert Scale: better than usual= 0, no more than usual= 1, worse than usual= 2, much worse than usual= 3. For the bimodal scale: better than usual= 0, no more than usual= 0, worse than usual= 1, much worse than usual= 1. Sum all items for a total score. Score range. Range is 0 -11 for bimodal response format. Interpretation of scores. Higher score indicates more fatigue. Self report scale
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-aminopirydine | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | 4.3 (1.4) | 3.3 (1.8)

11. Secondary Outcome: Walk
Description: Timed 25 Foot Walk Test (T25-FW). The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. TIME LIMIT PER TRIAL (2) 3 minutes (180 seconds) per trial.
Time Frame: 5-10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- 4-aminopyridine: 20 weeks administration of 4-aminopyridine. The mean dose provided to the patients was 0.63 ± 0.05 mg per kg of body weight.
- Placebo: Identical placebo tablet administered bid for 20 weeks
Arm/Group | 4-aminopyridine | Placebo
Number analyzed (Participants) | 11 | 10
seconds | 15.2 (13.3) | 10.4 (5.7)

12. Secondary Outcome: Number of Participants With Abnormal Studies
Description: Safety surveillance will be done every two weeks from the beginning of the study, intentionally searching for adverse events (AE). EEG (Diffuse or focal cerebral dysfunction through demonstration of background slowing or presence of epileptiform activity assessed by a neurophysiologist) and laboratory tests (Presence of values higher of the normal value established by local laboratory and related to the administration of treatments), blood and urine samples: creatinine, blood urea nitrogen, total cholesterol, triglycerides, total direct, and indirect bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, creatinine kinase, lactic acid dehydrogenase, amylase and lipase. A complete blood cell count with differentials and a routine urinalysis and urine culture also obtained at each visit, will be done before the patients take 40, 50 and 60 mg/day. The number of participants with abnormal studies were reported.
Time Frame: 22 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 4-aminopyridine Treatment: 4-aminopyridine is given as gelatin capsules containing 4-aminopyridine 10 mg and microcrystalline cellulose as the excipient. Each patient will take two capsules every 8 hours after meals, for a total of 8 capsules/day. The 4-aminopyridine dosage will increase 10 mg/4 weeks by substitution of placebo instead of 4-aminopyridine capsules; such that patients will receive from 40 to 60 mg. distribute in 6capsules/day throughout the study.
Arm/Group | 4-aminopyridine Treatment | Placebo
Number analyzed (Participants) | 11 | 10
Participants
  Number of participants with abnormal lab results | 1 | 0
  Number of participants with abnormal EEG | 0 | 0

ADVERSE EVENTS:
Time Frame: 22 weeks
Description: An adverse event (also referred to as an adverse experience) can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporarily associated with the use of a drug, without any judgment about causality or relationship to the drug. An adverse event can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.
Groups:
- 4-aminopyridine: 22 weeks administration of 4-aminopyridine. The mean dose provided to the patients was 0.63 ± 0.05 mg per kg of body weight.
Arm/Group | 4-aminopyridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 7/11 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4-aminopyridine (N=11) | Placebo (N=10)
Insominia (Psychiatric disorders) | 7 | 8
Headache (Nervous system disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 6 | 3
Vertigo (Nervous system disorders) | 6 | 3
Tremor in hands (Nervous system disorders) | 4 | 1
Mouth/tongue paresthesias (Nervous system disorders) | 4 | 2
Hand/feet paresthesias (Nervous system disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1
Blurred vision (Eye disorders) | 2 | 0
Global muscle tremor (Nervous system disorders) | 2 | 0
Irritability (Psychiatric disorders) | 2 | 4
Eye pain (Eye disorders) | 2 | 1
Tingling in feet (Nervous system disorders) | 1 | 2
Abnormal taste in mouth (Nervous system disorders) | 1 | 0
Hypersomnia (Psychiatric disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
As the sample size is very small, it is recommended to increase the number of patients. The heterogeneity in cognitive processes would imply a greater restriction criteria in the selection of patients to avoid the ceiling effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes